CLINICAL TRIAL: NCT00903903
Title: Computer-Assisted Quantification of the Synovial Perfusion in Patients With Arthritis Using Two-Dimensional and Three-Dimensional Power Doppler Ultrasonography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: The Institutional Review Board of Taichung Veterans General Hospital, Institutional Review Board
Other Study IDs: IRB TCVGH No:C09048
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Synovitis
Keywords: active synovitis
MeSH Terms: conditions — Synovitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: RA patients with at least one active synovitis
- 2: Non-RA patients with at least one active synovitis

SUMMARY:
The purpose of this study is to compare the data obtained by computer-aided quantification of the synovial perfusion in patients with arthritis using two-dimensional and three-dimensional power Doppler ultrasonography and the clinical data used to represent the degree of joint inflammation. Intra- and inter-observer reliability of this method will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* patients with at least one painful swollen peripheral joint observed by a rheumatologist, including:

  * shoulder joints
  * elbow joints
  * wrist joints
  * metacarpophalangeal (MCP) AND
  * proximal interphalangeal (PIP) joints of hands, ankle joints, subtalar joints, mid-tarsal joints, MTP and PIP joints of feet

Exclusion Criteria:

* patients with active infection
* patients with concurrent malignant disease
* patients with a history of traumatic, septic, or cystal arthritis
* previous joint surgery, or isotopic synovectomy within the past 12 months before the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Arthritis patients who visited the Rheumatology out patient clinic in Taichung Veterans General Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan